CLINICAL TRIAL: NCT04566003
Title: Phase 1 Evaluation Comparing Tau PET Radiotracers, [18F]GTP1 and [18F]PI-2620 or [18F]MK-6240 in Subjects With Normal Cognition or Prodromal to Moderate Alzheimer's Disease
Brief Title: Evaluation Comparing Tau PET Radiotracers, [18F]GTP1 and [18F]PI-2620 or [18F]MK-6240 in Subjects With Normal Cognition or Prodromal to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: GN42801
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Alzheimer Disease (AD)
MeSH Terms: conditions — Alzheimer Disease | interventions — (18F)GTP1; ((18)F)PI-2620

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- [18F]PI-2620 PET, then [18F]GTP1 PET (Experimental): Participants will undergo one [18F]PI-2620 PET imaging session, then one [18F]GTP1 PET imaging session. Prior to each session, participants will be administered a bolus intravenous injection of approximately 5 millicurie (mCi) of [18F]PI-2620 or 7mCi of [18F]GTP1.
  Interventions: Drug: [18F]GTP1; Drug: [18F]PI-2620
- [18F]GTP1 PET, then [18F]MK-6240 (Experimental): Participants will undergo one [18F]GTP1 PET imaging session, then one [18F]MK-6240 PET imaging session. Prior to each session, participants will be administered a bolus intravenous injection of approximately 5 millicurie (mCi) of [18 F]MK-6240 or 7mCi of [18F]GTP1.
  Interventions: Drug: [18F]GTP1; Drug: [18F]MK-6240

INTERVENTIONS:
Drug: [18F]GTP1 — Participants will receive a bolus IV of approximately 7mCi of [18F]GTP1 radiotracer.
Drug: [18F]PI-2620 — Participants will receive a bolus IV of approximately 5mCi of [18F]PI-2620 radiotracer.
  Arms: [18F]PI-2620 PET, then [18F]GTP1 PET
Drug: [18F]MK-6240 — Participants will receive a bolus IV of approximately 5mCi of [18F]MK-6240 radiotracer.
  Arms: [18F]GTP1 PET, then [18F]MK-6240

SUMMARY:
The study aims to compare tau targeted radiotracers [18F]GTP1 and [18F]PI-2620 or [18F]MK-6240 in subjects with normal cognition or prodromal to moderate Alzheimer's disease (AD).

ELIGIBILITY:
Inclusion Criteria

* Cognitively normal subjects aged 65 to 90 years and prodromal to mild AD subjects aged 50 to 90 years, inclusive at the time of screening.
* Prodromal to moderate AD subjects: Meet the National Institute on Aging - Alzheimer's Association (NIA-AA) core clinical criteria for mild cognitive impairment (MCI) due to AD, probable AD dementia or AD dementia
* Have a Clinical Dementia Rating (CDR) score of 0 (cognitively normal) or 0.5 (prodromal to moderate AD) at screening
* Have an Mini-Mental State Examination (MMSE) score 10-30 inclusive
* Have Aβ PET imaging demonstrating Aβ binding based on qualitative visual read at screening or using an acceptable historical PET scan (cognitively normal subjects will be assessed with Aβ PET at screening but will not be required to demonstrate Aβ binding).
* A brain MRI consistent with normal cognition or that supports a diagnosis of prodromal to moderate AD, with no evidence of other significant neurologic pathology. A previously acquired research MRI within the last 12 months may be used if deemed acceptable by the investigator and no significant clinically relevant changes have occurred since the prior MRI was obtained
* The subject has an appropriate study partner capable of participating in CDR assessment and, if necessary, of accompanying the subject
* For cognitively normal subjects only: History of at least one first degree relative with diagnosis of Alzheimer's disease (self-reported by the potential subject and/or confirmed by the study partner).

Exclusion Criteria

* Current or prior history of any alcohol or drug abuse within the last 2 years
* Prior participation in other research protocols or clinical care in the last year in addition to the radiation exposure expected from participation in this clinical study, such that radiation exposure exceeds the effective dose of 50 millisievert (mSv), which would be above the acceptable annual limit established by the US Federal Guidelines
* Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease
* MRI evidence of cerebrovascular disease, infectious disease, space-occupying lesions, normal pressure hydrocephalus, or other central nervous system (CNS) disease
* Implants that have not been certified for MRI or history of claustrophobia in MRI, unless an acceptable previously acquired research MRI is available

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to approximately 4 days after administration of each radiotracer
Brain tau burden as measured by [18F]PI-2620 - PET | Approximately 1 hour after injection of [18F]PI-2620
Brain tau burden as measured by [18F]GTP1 - PET | Approximately 1 hour after injection of [18F]PI-2620
Brain tau burden as measured by [18F]MK-6240 - PET | Approximately 1 hour after injection of [18F]MK-6240

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Invicro, a Konica Minolta company, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).